CLINICAL TRIAL: NCT04204421
Title: The Experience Sampling Method (ESM): Validation of a Newly Developed Real-time Patient-Reported Outcome Measure (PROM) and Its Evaluation of Triggers for Functional Dyspepsia
Brief Title: ESM in Functional Dyspepsia
Acronym: MEASuRE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METC 19-077 / NL71810.068.19
Record Dates: First submitted 2019-12-09; First posted 2019-12-19 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Dyspepsia; Dyspepsia and Other Specified Disorders of Function of Stomach
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experience Sampling Method (ESM) (Experimental): Both patients with functional dyspepsia and healthy controls will be asked to fill out ESM questionnaires during 1 week. Moreover, at the end of this week, usual questionnaires for complaints assessment will be filled out.
  Interventions: Other: Experience Sampling Method (ESM)

INTERVENTIONS:
Other: Experience Sampling Method (ESM) — Experience Sampling Method (ESM) is a method for real time complaints assessment where people are asked to fill out a questionnaire 10 times per day at random moments. This will be done via a mobile phone application.
  Other Names: ESM

SUMMARY:
Background:

Reliable patient reported outcome measures (PROM's) for symptom assessment in functional dyspepsia (FD) are essential in order to evaluate dyspeptic symptoms, identify potential symptom triggers and optimize therapeutic strategies, since biological markers are unavailable. Currently used symptom assessment methods, i.e. end-of-day or end-of-week questionnaires, have considerable limitations. The Experience Sampling Method (ESM), an electronic questioning method characterized by random and repeated, momentary assessments in the subject's current state and environment, might overcome these limitations. The aim of this study is to assess the validity and reliability of an FD-specific electronic patient-reported outcome measure (ePRO), based on the Experience Sampling Method-principle, for symptom assessment and identification of symptom triggers in patients with functional dyspepsia.

Objective:

The aim of this study is to assess the validity and reliability of an FD-specific electronic patient-reported outcome measure (ePRO), based on the Experience Sampling Method-principle, for symptom assessment and identification of symptom triggers in patients with functional dyspepsia. In order to measure this, internal consistency, test-retest reliability, concurrent validity and the accuracy to differentiate between dyspeptic patients and healthy controls of the developed ePRO will be assessed. In addition, to objectify specific triggers for the onset of gastrointestinal symptoms in dyspepsia, using the FD-specific ESM tool.

ELIGIBILITY:
Both patients with functional dyspepsia (36) as healthy controls (36) will be included

Inclusion Criteria for patients with functional dyspepsia:

• A diagnosis of functional dyspepsia according to ROME IV criteria (2):

* One or more of the following:
* Bothersome postprandial fullness
* Bothersome early satiation
* Bothersome epigastric pain
* Bothersome epigastric burning

AND

* No evidence of structural disease (confirmed by upper endoscopy) that is likely to explain the symptoms.
* Criteria fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.

  * Age between 18 and 75 years;
  * Ability to understand and speak the Dutch language;
  * Ability to understand how to utilize the ESM tool.

Inclusion criteria for healthy volunteers:

* Age between 18 and 75 years
* Ability to understand and speak the Dutch language
* Ability to understand how to utilize the ESM tool.

Exclusion Criteria for patients with functional dyspepsia:

* Any organic explanation for the gastrointestinal complaints;
* Initiation of regularly used medication from one month before inclusion until the end of study participation;
* A history of upper digestive surgery influencing end points
* A history of radiation therapy of the abdomen
* Pregnancy

Exclusion Criteria for healthy controls:

* Current diagnosis of any gastrointestinal disorder
* Current gastrointestinal symptoms suiting the ROME IV criteria for FD
* Initiation of regularly used medication from one month before inclusion until the end of study participation
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in experience sampling method (ESM) scores | 10 times daily, during 1 week
  Using the MEASuRE-D app, the same ESM questionnaire will be filled in 10 times per day at random intervals. This results in a lot of real-time data on patient symptom scores on which changes over the course of the day can be seen.
Patient complaint diary | End of day 1, end of day 2, end of day 3, end of day 4, end of day 5, end of day 6, end of day 7
  Using the MEASuRE-D app, patients will fill out a complaints diary at the end of each day during 7 days

SECONDARY OUTCOMES:
Questionnaire for demographic characteristics | On day 7
  A questionnaire for demographic characteristics will be filled in by participants.
PAGI-SYM questionnaire | On day 7
  the Patient Assessment of Upper Gastrointestinal Disorders Symptom Severity index (PAGI-SYM) questionnaire will be filled in by participants. Questions about upper gastrointestinal symptoms are asked on a 6 point likert scale with 0 indicating not at all and 5 indicating very severe.
NDI questionnaire | On day 7
  The Nepean Dyspepsia Index (NDI) questionnaire will be filled in by participants. The NDI questionaire consists of various questions.
  Questions about the effects of upper gastrointestinal symptoms are asked on a 5 point likert scale with 1 indicating not at all/almost never and 5 indicating very severe/always.
GSRS questionnaire | On day 7
  The Gastrointestinal Symptom Rating Scale (GSRS) will be filled in by participants. Questions about gastrointestinal symptoms are asked on a 7 point likert scale with 0 indicating not at all and 6 indicating very severe.
PHQ-9 questionnaire | On day 7
  The Patient Health Questionnaire-9 (PHQ-9) will be filled in by participants. Questions about the severity of depressive symptoms are asked on a scale from 0 - 3, where 0 indicates not at all, 1 indicates some days, 2 indicates more than half of the days, and 3 indicates almost every day.
GAD-7 questionnaire | On day 7
  The Generalized Anxiety Disorder-7 (GAD-7) questionnaire will be filled in by participants. Questions about the severity of anxiety symptoms are asked on a scale from 0 - 3, where 0 indicates not at all, 1 indicates some days, 2 indicates more than half of the days, and 3 indicates almost every day.
PHQ-15 questionnaire | On day 7
  The Patient Health Questionnaire-15 (PHQ-15) will be filled in by participants. Questions about somatization symptoms are asked in the following matter: how often have you been bothered by "..." on a scale from 0 - 2, where 0 indicates not at all, 1 indicates bothered a little, and 2 indicates bothered a lot.
SF-36 questionnaire | On day 7
  The Short Form-36 (SF-36) questionnaire will be filled in by participants and consits of various types of questions.
  Some questions about how their health limits them in certain daily activities are asked on a scale of 1-3, with 1 indicating limits severely, 2 indicating limits a little, and 3 indicating not limited at all Some questions about problems in participants' work or daily activities due to physical health, emotional problems are dichotomous with 1 indicating yes and 2 indicating no Some questions about how participants felt themselves during a period are asked on a 6 point scale with 1 indicating all the time, 2 indicating most of the time, 3 indicating often, 4 indicating sometimes, 5 indicating occasionally, and 6 indicating not at all Participants need to indicate how much a few statements apply to them with 1 indicating completely correct, 2 indicating mostly correct, 3 indicating I don't know, 4 indicating mostly incorrect, and 5 indicating completely correct

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Masclee, Prof., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klaassen T, Vork L, Smeets FGM, Troost FJ, Kruimel JW, Leue C, Masclee AAM, Keszthelyi D. The Interplay Between Stress and Fullness in Patients With Functional Dyspepsia and Healthy Controls: An Exploratory Experience Sampling Method Study. Psychosom Med. 2022 Apr 1;84(3):306-312. doi: 10.1097/PSY.0000000000001012. PMID 34524263